CLINICAL TRIAL: NCT02776865
Title: Does Ultrasound-guided Suprascapular Nerve Block Provide Additional Benefit
Brief Title: Does Ultrasound-guided Suprascapular Nerve Block Provide Additional Benefit Over Traditional Rehabilitation Program for Patients With Chronic Shoulder Pain
Acronym: 2015/8/1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015-09-009C
Record Dates: First submitted 2016-05-16; First posted 2016-05-18 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-03

CONDITIONS: Suprascapular Nerve Block
Keywords: suprascapular nerve block
MeSH Terms: interventions — Lidocaine; Physical Therapy Modalities; Rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- physical therapy and suprascapular nerve block (Experimental): patient received ultrasound-guided suprascapular nerve block as well as physical therapy.
  Interventions: Drug: suprascapular nerve block; Other: physical therapy
- physical therapy only (Active Comparator): patient received physical therapy only.
  Interventions: Other: physical therapy

INTERVENTIONS:
Drug: suprascapular nerve block — 4ml 2% xylocaine
  Other Names: 4cc 2% xylocaine
  Arms: physical therapy and suprascapular nerve block
Other: physical therapy — patient received traditional physical therapy, including therapeutic exercise and stretch exercise
  Other Names: rehabilitation

SUMMARY:
This study was conducted to compare the efficacy of hydrodilatation with hyaluronic acid under ultrasonographic guidance plus physical therapy (PT) with that of PT alone for treating adhesive capsulitis

ELIGIBILITY:
Inclusion Criteria:

1. chronic shoulder pain with duration of complaints more than 3 months
2. diagnosis of frozen shoulder or rotator cuff disorder

Exclusion Criteria:

1. other conditions involving the shoulder ( rheumatoid arthritis, Hill-Sachs lesions,osteoporosis, or malignancies in the shoulder region);
2. neurologic deficits affecting shoulder function in normal daily activities;
3. shoulder pain caused by cervical radiculopathy
4. a history of drug allergy to xylocaine
5. pregnancy or lactation;
6. received injection into the affected shoulder during the preceding 3 months

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
change in constant shoulder score | at 4, 12 wk
  the total constant score ranges from 0 to 100 points, with higher scores indicative of better function. The score is divided into four sections: pain, activity of daily living, ROM and strength

SECONDARY OUTCOMES:
change in pain intensity | at 4, 12 wk
  pain intensity was measured by visual analog scale.
change in Shoulder Pain And disability index | at 6, 12 wk
  The Shoulder Pain and Disability Index (SPADI) is a self-administered questionnaire that consists of two dimensions, one for pain and the other for functional activities. The pain dimension consists of five questions regarding the severity of an individual's pain. Functional activities are assessed with eight questions designed to measure the degree of difficulty an individual has with various activities of daily living that require upper-extremity use. The SPADI takes 5 to 10 minutes for a patient to complete and is the only reliable and valid region-specific measure for the shoulder.
change in glenohumeral joint range of motion | at 4, 12 wk
  Shoulder flexion, abduction, external rotation and internal rotation were measured with goniometer with patient in supine position.

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei veteran general hospital, Taipei, Taiwan